CLINICAL TRIAL: NCT05358938
Title: Exercise to Boost Response to Checkpoint Blockade Immunotherapy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20854
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Melanoma; Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma
Keywords: Exercise; Checkpoint Blockade Immunotherapy; Immunotherapy; Skin Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Motor Activity; Skin Neoplasms | interventions — Exercise; Immune Checkpoint Inhibitors; avelumab; cemiplimab; Ipilimumab; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Adjuvant Arm with Exercise (Experimental): Participants will receive clinical care following Moffitt standards for the patient's disease type and therapeutic setting. Adjuvant participants will receive 1 year [currently 9-18 cycles] of therapy with avelumab, cemiplimab, ipilimumab, nivolumab, pembrolizumab or relatlimab, or currently approved standard of care treatment, either alone or in combination. Participants also will complete 30 minutes of moderate exercise on an arm ergometer, a cycle ergometer, or a treadmill prior to each administration of standard of care checkpoint blockade immunotherapy across all cycles. Blood samples will be collected at 1) baseline (upon arrival to clinic), 2) post-exercise, and 3) post-infusion. Blood samples will be obtained on the first, third, midpoint, and final infusion dates.
  Interventions: Other: Exercise; Drug: Checkpoint Blockade, Immune
- Adjuvant Arm without Exercise (Active Comparator): Participants will receive clinical care following Moffitt standards for the patients disease type and therapeutic setting. Adjuvant participants will receive one year [currently 9-18 cycles] of therapy with avelumab, cemiplimab, ipilimumab, nivolumab, pembrolizumab, relatlimab, or currently approved standard of care treatment, either alone or in combination. Blood samples will be collected at 1) baseline (upon arrival to clinic) and 2) post-infusion. Blood samples will be obtained on the first, third, midpoint, and final infusion dates.
  Interventions: Drug: Checkpoint Blockade, Immune
- Neoadjuvant Arm with Exercise (Experimental): Participants will complete 30 minutes of moderate exercise on an arm ergometer, a cycle ergometer, or a treadmill prior to each administration of standard of care checkpoint blockade immunotherapy across all cycles. Neoadjuvant participants will receive up to 4 cycles of therapy with avelumab, cemiplimab, ipilimumab, nivolumab, pembrolizumab, or relatlimab, or currently approved standard of care treatment, either alone or in combination. Blood samples will be collected at 1) baseline (upon arrival to clinic), 2) post-exercise, and 3) post-infusion. Blood samples will be obtained on the first and third infusion dates.
  Interventions: Other: Exercise; Drug: Checkpoint Blockade, Immune
- Neoadjuvant Arm without Exercise (Active Comparator): Participants will receive clinical care following Moffitt standards for the patient's disease type and therapeutic setting. Neoadjuvant participants will receive up to 4 cycles of therapy with avelumab, cemiplimab, ipilimumab, nivolumab, pembrolizumab, or relatlimab, or currently approved standard of care treatment, either alone or in combination. Participants also will complete 30 minutes of moderate exercise on an arm ergometer, a cycle ergometer, or a treadmill prior to each administration of standard of care checkpoint blockade immunotherapy across all cycles. Blood samples will be collected at 1) baseline (upon arrival to clinic), 2) post-exercise, and 3) post-infusion. Blood samples will be obtained on the first and third infusion dates.
  Interventions: Drug: Checkpoint Blockade, Immune

INTERVENTIONS:
Other: Exercise — 30 minutes of moderate exercise on an arm ergometer, a cycle ergometer, or a treadmill prior to each administration of standard of care checkpoint blockade immunotherapy across all cycles
  Arms: Adjuvant Arm with Exercise; Neoadjuvant Arm with Exercise
Drug: Checkpoint Blockade, Immune — Participants will receive clinical care following Moffitt standards for the patient's disease type and therapeutic setting.
  Other Names: Avelumab; Cemiplimab; Ipilimumab; Nivolumab; Pembrolizumab

SUMMARY:
30 minutes of moderate exercise on an arm ergometer, a cycle ergometer, or a treadmill prior to each administration of standard of care checkpoint blockade immunotherapy across all cycles

ELIGIBILITY:
* Inclusion Criteria:
* Age ≥ 18 years
* Able to read and speak English fluently
* Capable of giving informed consent
* Reported ability to complete 20-30 minutes moderate exercise per positive response to "can you currently walk unaided for six minutes or more?".
* Scheduled for first-time checkpoint blockade immunotherapy with FDA-approved drugs, including avelumab, cemiplimab, ipilimumab, nivolumab, pembrolizumab or relatlimab in the absence of other therapies (e.g. targeted therapy)
* Melanoma patients (adjuvant setting)
* Melanoma patients (neoadjuvant setting)
* cuSCC patients (neoadjuvant setting)
* Merkel cell carcinoma patients (neoadjuvant setting)

Participants may also be required to have a full COVID vaccination series; the most up-to-date best practice guidelines for research at Moffitt Cancer Center will dictate the need for such a vaccination series.

Exclusion Criteria:

* Presence of medical conditions, such as severe cardiovascular disease for which an exercise intervention may not be warranted.
* Presence of major postoperative complications for which an exercise intervention may not be warranted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Participants Consenting to Trial | Up to 12 months
  Proportion of patients approached who consent to participate in study, and investigators will determine the 95% confidence interval
Participants Completing Exercise | Up to 12 months
  Proportion of participants randomized to the exercise intervention who complete at least 75% of schedule exercise routines; 95% CI will be determined for this proportion.
Impact of Exercise on Tumor Immunological Biomarkers - Adjuvant Setting | Up to 12 Months
  The length of time without signs or symptoms of cancer
Pathological Complete Response (pCR) - Neoadjuvant Setting | Up to 4 Months
  The occurrence of pathological complete response in resected tumor tissue. pCR will be determined by absence of tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kanetsky, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE